CLINICAL TRIAL: NCT03223415
Title: Effectiveness of Isolating Clostridium Difficile Asymptomatic Carriers on the Incidence of Infections; A Cluster Randomized Feasibility Trial
Brief Title: Effectiveness of Isolating Clostridium Difficile Asymptomatic Carriers on the Incidence of Infections
Acronym: EFFICACI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yves Longtin (Other)
Collaborators: Becton, Dickinson and Company (Industry); Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Sponsor-Investigator, Yves Longtin, Chair, Infection Prevention and Control Unit, Jewish General Hospital
Organization: Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MM-CODIM-MBM-16-264; BDS-MCDIF04 (Other: Becton, Dickinson and Company)
Record Dates: First submitted 2017-05-25; First posted 2017-07-21 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile infection; Infection Control; Prevention; Asymptomatic carriage; Colonization; Pilot Study; Contact Precaution; Detection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Detection and isolation of C. difficile carriers
  Interventions: Other: Detection and isolation of C. difficile carriers
- Control arm (No Intervention): No detection of C. difficile carriers upon admission and no implementation of contact isolation precautions for C. difficile carriers

INTERVENTIONS:
Other: Detection and isolation of C. difficile carriers — Screening for C. difficile carriage will be conducted by performing a polymerase chain reaction (PCR) assay detecting the toxin B gene (tcdB) on a rectal swab. Screening will occur within 24 h of admission to the ward. To ensure compliance with the policy, automatic orders will be developed. The patient care nurse will perform the screenings. The results will be reported according to the standard institutional policy.
  Isolation precautions for C. difficile carriers: healthcare workers will also follow a set of isolation precaution rules during the care of C. difficile carriers. C. difficile carriers will remain under isolation precaution as long as they remain carriers and on the intervention ward. Precautions would be discontinued upon discharge from the ward.
  Arms: Experimental arm

SUMMARY:
Background: There is an urgent need to develop new strategies to prevent Clostridium difficile infections (CDI). A recent study suggests that a novel infection control bundle (IC bundle) can lead to a significant decrease in the incidence of CDI in acute-care hospitals. This IC bundle consists in screening patients for C. difficile carriage upon their admission combined with implementation of isolation precautions for carriers. Further investigations are required to confirm these findings.

Objective: To evaluate the feasibility of implementing a multicenter interventional study to further to investigate the efficacy of this IC bundle.

Methods: Prospective, cluster randomized feasibility trial of 2 infection control strategies (a "standard" and an "experimental" strategy) to reduce transmission of C. difficile among patients in 20 medical wards in 5 acute-care facilities in Quebec. Wards will be randomized (1:1) to one of the 2 interventions. Each intervention will be applied to all patients present on selected wards. The study will be divided into (1) a 3-month baseline period; (2) a 2-week randomization and implementation period; and (3) an 8-week intervention period.

Intervention: The "experimental strategy" includes the components of the above-mentioned IC bundle. The "standard strategy" will not implement the IC bundle.

Outcomes: As a feasibility study, process evaluation will form the primary and secondary outcomes. These outcomes will allow to determine whether a future main trial is possible and desirable.

Hypothesis: We hypothesize that the intervention will be implementable across the study wards.

Significance: This study is essential to plan a subsequent definitive trial to determine whether the IC bundle can prevent CDI.

DETAILED DESCRIPTION:
C. difficile is a gram-negative anaerobic bacteria that causes C. difficile infection (CDI), a disease involving the colon and causing symptoms ranging from mild diarrhea to fulminant colitis. C. difficile can spread from patients to patients in acute-care hospitals. Transmission is believed to occur mainly from patients with active disease, but patients who carry the bacteria without any symptom (called C. difficile carriers) can also transmit the bacteria to other patients.

Preliminary evidence that suggest that detecting C. difficile carriers to place them under isolation precautions can lead to a decrease in the incidence of CDI. In order to investigate this question, large-scale clinical trials will be ultimately required. In order to plan such large-scale study, there is a need to perform a preliminary feasibility trial. The current study will assess the feasibility, acceptability and logistical considerations of implementing a multicenter intervention consisting of the detection and isolation of C. difficile carriers on hospital admission, in order to guide the design of a definitive trial. This objective is essential considering the paucity of published data on this topic.

ELIGIBILITY:
Because both strategies will be applied at the ward level, the inclusion and exclusion criteria apply to wards, not to individual patients. All patients and healthcare workers on each ward will be assigned to the intervention.

Inclusion criteria:

Clusters (i.e. wards) are eligible to take part in the study if they meet the following criteria:

* Adult medical or surgical wards;
* Patient volume: ≥5 admissions/month and ≥600 patient days/month in 2015;
* Incidence rate of CDI of ≥5/10 000 patient-days based during in 2014-2015;
* Commitment by the hospital administration to have the hospital undergo randomization for the trial (Willingness to be randomized in either arm of the study);
* Institutional agreement to screen all eligible new admissions for CD carriers and isolate CD carriers in accordance with the study protocol;
* Signed protocol signature page indicating willingness to enroll the ward in the study from the director of the hospital;
* Capacity to implement protocol (screening, isolation, respect of contact precautions);
* Capacity to screen patients by PCR with a turnaround time of <24 h;
* Participation in the Quebec CDI surveillance program (SPIN-CD);
* No existing protocol to detect and isolate CD carriers (isolation of CDI patients with resolved diarrhea allowed);
* Stable use of infection-prevention initiatives and products during the baseline period;
* Agreement to refrain from adopting new initiatives that would conflict with the trial.

Exclusion criteria:

* Wards planning to enroll subjects in other studies that aim to eradicate or prevent colonization with C. difficile or management strategies that have CD carriers or CDI as an outcome.
* Gender-biased wards (gynecology/ obstetrics, urology).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4138 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Rate of admission screening for C. difficile carriage | 8 weeks
  Rate of admission screening for C. difficile carriage, defined as the number of patients who were screened on admission divided by the number of admitted patients per 4-week period

SECONDARY OUTCOMES:
Healthcare worker compliance with the isolation precautions | 8 weeks
  Healthcare worker compliance with the isolation precautions, defined as the number of opportunities in which healthcare workers complied with the isolation precaution upon entering the room of a C. difficile carrier divided by the total number of healthcare workers who entered the room.
Rate of rejection of screening assays | 8 weeks
  Rate of rejection of rectal swabs, defined as the number of rectal swabs submitted to the laboratory for C. difficile screening assay that were rejected for any reason divided by the total number of rectal swabs submitted for C. difficile screening assay per 4-week period.
Healthcare worker compliance with hand washing | 8 weeks
  Healthcare worker compliance with hand washing, defined as the number of opportunities in which healthcare workers complied with the hand washing policy upon exiting the room of a C. difficile carrier divided by the total number of hand washing opportunities upon exiting the room of a C. difficile carrier.
Proportion of screening assays with proper turnaround time | 8 weeks
  Proportion of screening assays with proper turnaround time, defined as the number of screening samples with a < 24 hour turnaround time (TAT) divided by the number of screening samples submitted to the laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Longtin, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (5):
- Canada (5):
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Centre Hospitalier Sainte-Marie, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Longtin Y, Paquet-Bolduc B, Gilca R, Garenc C, Fortin E, Longtin J, Trottier S, Gervais P, Roussy JF, Levesque S, Ben-David D, Cloutier I, Loo VG. Effect of Detecting and Isolating Clostridium difficile Carriers at Hospital Admission on the Incidence of C difficile Infections: A Quasi-Experimental Controlled Study. JAMA Intern Med. 2016 Jun 1;176(6):796-804. doi: 10.1001/jamainternmed.2016.0177. PMID 27111806